CLINICAL TRIAL: NCT05948215
Title: Jing Si Herbal Tea in the Treatment of Dyspeptic Symptoms and Psychophysical Burden in Patients With Functional dyspepsia--a Double-blind, Randomized, Placebo-controlled Study
Brief Title: Jing Si Herbal Tea in the Treatment of Dyspeptic Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB110-232-A
Record Dates: First submitted 2023-07-05; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-06

CONDITIONS: Functional Gastrointestinal Disorders; Healthy Subjects
Keywords: Jing Si Herbal Tea Liquid Packet; psychophysical burden
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jing Si Herbal Tea Liquid Packet (Experimental): Participants received Jing Si Herbal Tea Liquid Packet 15 mg tablet orally once daily for 28 days.
  Interventions: Dietary Supplement: Jing Si Herbal Tea Liquid Packet
- Jing Si Herbal Tea Liquid Packet Placebo (Placebo Comparator): Participants received Jing Si Herbal Tea Liquid Packet Placebo 15 mg tablet orally once daily for 28 days.
  Interventions: Dietary Supplement: Jing Si Herbal Tea Liquid Packet Placebo

INTERVENTIONS:
Dietary Supplement: Jing Si Herbal Tea Liquid Packet — The preliminary data demonstrated that the Jing Si Herbal Tea Liquid Packet may improve gastrointestinal symptoms and anxiety in patients with Coronavirus disease 2019(COVID-19). Therefore,this study aims to investigate the impact of the Jing Si Herbal Tea Liquid Packet on psychophysical burden and metabolites of microbiota in patients with FD through a double-blind randomized manner.
  Arms: Jing Si Herbal Tea Liquid Packet
Dietary Supplement: Jing Si Herbal Tea Liquid Packet Placebo — Compared with the improvement effect of Jing Si Herbal Tea Liquid Packet, to avoid participants thinking that the improvement is due to psychological effects.
  Other Names: Placebo
  Arms: Jing Si Herbal Tea Liquid Packet Placebo

SUMMARY:
Dyspepsia refers to chronic or recurrent upper gastrointestinal symptoms. According to the Rome IV criteria, functional dyspepsia (FD) symptoms included meal-related fullness, early satiation, epigastric pain or burning which are unexplained after routine investigation. FD causes substantial psychophysical burden because of its unknown etiology and high prevalence. Although FD is currently associated with local inflammation of the gastrointestinal tract and microbiota alteration, current available treatments for FD are of limited effectiveness. In view of this, many studies have applied Chinese herbal medicine in FD and achieved some therapeutic benefit. The Jing Si Herbal Tea composed of eight native Taiwanese herbs (wormwood, hickory grass, Ophiopogon japonicus, houttuynia cordata, platycodon, licorice, perilla leaves, chrysanthemum) has obtained a special export license from the Ministry of Health and Welfare. The Jing Si Herbal Tea also has been registered in clinical trials as a complementary treatment for COVID-19. The preliminary data demonstrated that the Jing Si Herbal Tea may improve gastrointestinal symptoms and anxiety in patients with COVID-19. Therefore, this study aims to investigate the impact of the Jing Si Herbal Tea on psychophysical burden and metabolites of microbiota in patients with FD through a double-blind randomized manner.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-79 years old.
2. Those who meet the definition of functional dyspepsia (FD). (Functional dyspepsia (FD) is chronic (once a week, lasting at least three months, at least six months before the first symptom) upper gastrointestinal symptoms (any of the following): postprandial abdominal distension, easy to feel full, Epigastric pain or burning sensation in the upper abdomen, and no symptoms of gastrointestinal bleeding or significant weight loss, no abnormality after upper gastrointestinal endoscopy).
3. Be conscious and willing to sign the subject's consent form.

Exclusion Criteria:

1. Abnormal liver and kidney function;
2. Abnormal blood tests and thyroid abnormalities;
3. Have received surgery on the digestive tract;
4. Abnormal upper gastrointestinal endoscopy;
5. Have gastric pylori infection;
6. Antibiotics are being used for infectious diseases;
7. Pregnant or breastfeeding women;
8. Suffering from heart, liver, or kidney failure;
9. Physical weakness, allergies, coldness, chronic diseases, poor kidney function, infants under three years old, children, Pregnancy, lactation, menstrual period.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Pain on the Visual Analogue Scale (VAS) at day 28 | Baseline and day 28
  Possible scores range from 0 (No pain) to 10 (Worst possible pain) Change = (day 28 Score - Baseline Score).
Change from Baseline on the Pittsburgh sleep quality index (PSQI) at day 28 | Baseline and day 28
  Possible scores range from 0 (Never) to 3 (Occurs three times a week times or more) 0=Never 1=Less than once a week 2=Occurs once or twice a week 3=Occurs three times a week times or more Change = (day 28 Score - Baseline Score).
Change from Baseline on the Taiwanese Depression Scale (TDQ) at day 28 | Baseline and day 28
  Possible scores range from 0 (Never) to 3 (Always) 0=Never 1=Sometimes 2=Often 3=Always Change = (day 28 Score - Baseline Score).
Change from Baseline on the State-Trait Anxiety Inventory (STAI) at day 28 | Baseline and day 28
  Possible scores range from 1 (Never) to 4 (Always)
  1=Never 2=Sometimes 3=Often 4=Always Change = (day 28 Score - Baseline Score).
Change from Baseline on the Perceived Stress Scale(PSS-10) at day 28 | Baseline and day 28
  Possible scores range from 0 (Never) to 4 (Always) 0=Never 1=Rarely 2=Sometimes 3=Often 4=Always Change = (day 28 Score - Baseline Score).
Change from Baseline on the Patient Assessment of Upper Gastrointestinal Symptoms(PAGI-SYM) at day 28 | Baseline and day 28
  Possible scores range from 0 (No pain) to 5 (Very serious) 0=No pain 1=Very slightly 2=Slight 3=About medium 4=Serious 5=Very serious Change = (day 28 Score - Baseline Score).

CONTACTS AND LOCATIONS:
Locations (1):
- Hualien Tzu Chi Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sperber AD, Bangdiwala SI, Drossman DA, Ghoshal UC, Simren M, Tack J, Whitehead WE, Dumitrascu DL, Fang X, Fukudo S, Kellow J, Okeke E, Quigley EMM, Schmulson M, Whorwell P, Archampong T, Adibi P, Andresen V, Benninga MA, Bonaz B, Bor S, Fernandez LB, Choi SC, Corazziari ES, Francisconi C, Hani A, Lazebnik L, Lee YY, Mulak A, Rahman MM, Santos J, Setshedi M, Syam AF, Vanner S, Wong RK, Lopez-Colombo A, Costa V, Dickman R, Kanazawa M, Keshteli AH, Khatun R, Maleki I, Poitras P, Pratap N, Stefanyuk O, Thomson S, Zeevenhooven J, Palsson OS. Worldwide Prevalence and Burden of Functional Gastrointestinal Disorders, Results of Rome Foundation Global Study. Gastroenterology. 2021 Jan;160(1):99-114.e3. doi: 10.1053/j.gastro.2020.04.014. Epub 2020 Apr 12. PMID 32294476
- [Result] Stanghellini V, Chan FK, Hasler WL, Malagelada JR, Suzuki H, Tack J, Talley NJ. Gastroduodenal Disorders. Gastroenterology. 2016 May;150(6):1380-92. doi: 10.1053/j.gastro.2016.02.011. PMID 27147122
- [Result] Talley NJ, Ford AC. Functional Dyspepsia. N Engl J Med. 2015 Nov 5;373(19):1853-63. doi: 10.1056/NEJMra1501505. No abstract available. PMID 26535514
- [Result] Wauters L, Talley NJ, Walker MM, Tack J, Vanuytsel T. Novel concepts in the pathophysiology and treatment of functional dyspepsia. Gut. 2020 Mar;69(3):591-600. doi: 10.1136/gutjnl-2019-318536. Epub 2019 Nov 29. PMID 31784469
- [Result] Gwee KA, Holtmann G, Tack J, Suzuki H, Liu J, Xiao Y, Chen MH, Hou X, Wu DC, Toh C, Lu F, Tang XD. Herbal medicines in functional dyspepsia-Untapped opportunities not without risks. Neurogastroenterol Motil. 2021 Feb;33(2):e14044. doi: 10.1111/nmo.14044. Epub 2020 Nov 30. PMID 33258198
- [Result] Masuy I, Van Oudenhove L, Tack J. Review article: treatment options for functional dyspepsia. Aliment Pharmacol Ther. 2019 May;49(9):1134-1172. doi: 10.1111/apt.15191. Epub 2019 Mar 28. PMID 30924176
- [Result] Ford AC, Moayyedi P, Black CJ, Yuan Y, Veettil SK, Mahadeva S, Kengkla K, Chaiyakunapruk N, Lee YY. Systematic review and network meta-analysis: efficacy of drugs for functional dyspepsia. Aliment Pharmacol Ther. 2021 Jan;53(1):8-21. doi: 10.1111/apt.16072. Epub 2020 Sep 16. PMID 32936964
- [Result] Teschke R, Wolff A, Frenzel C, Eickhoff A, Schulze J. Herbal traditional Chinese medicine and its evidence base in gastrointestinal disorders. World J Gastroenterol. 2015 Apr 21;21(15):4466-90. doi: 10.3748/wjg.v21.i15.4466. PMID 25914456
- [Result] Suzuki H, Matsuzaki J, Fukushima Y, Suzaki F, Kasugai K, Nishizawa T, Naito Y, Hayakawa T, Kamiya T, Andoh T, Yoshida H, Tokura Y, Nagata H, Kobayakawa M, Mori M, Kato K, Hosoda H, Takebayashi T, Miura S, Uemura N, Joh T, Hibi T, Tack J; Rikkunshito study group. Randomized clinical trial: rikkunshito in the treatment of functional dyspepsia--a multicenter, double-blind, randomized, placebo-controlled study. Neurogastroenterol Motil. 2014 Jul;26(7):950-61. doi: 10.1111/nmo.12348. Epub 2014 Apr 28. PMID 24766295
- [Result] Drossman DA. Functional Gastrointestinal Disorders: History, Pathophysiology, Clinical Features and Rome IV. Gastroenterology. 2016 Feb 19:S0016-5085(16)00223-7. doi: 10.1053/j.gastro.2016.02.032. Online ahead of print. PMID 27144617

DOCUMENTS (2):
  • Study Protocol (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/15/NCT05948215/Prot_000.pdf
  • Informed Consent Form (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/15/NCT05948215/ICF_001.pdf